CLINICAL TRIAL: NCT04966104
Title: ODYSSEE-vCHAT Pilot Trial: a Virtual Community Promoting Health Literacy, Self-Care, and Peer Support for Heart Failure
Brief Title: ODYSSEE-vCHAT Pilot Trial for Heart Failure
Acronym: ODYSSEE-vCHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-5960; PJT173222 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); 5117 (Other: Sunnybrook Hospital Research Ethics Board); 21-022-E (Other: Mount Sinai Hospital Research Ethics Board)
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
Keywords: Digital health; Digital counselling; Self-care; Clinical trial; Clinical outcomes; Cognitive-behavioural therapy; Health-related quality of life; Motivational interviewing; eHealth; Social Networking
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Double arm, parallel group, single-blind randomized trial
Who Masked: Investigator
Masking Description: An independent statistician logged on to a secure program (managed by the UHN THETA institute) that used randomly permuted blocks to assign subjects to ODYSSEE-vCHAT or the control group. To reduce the chance of patient allocation being predictable, we followed the convention whereby the block sizes and the fraction of each block size were known only by an independent statistician. We tested this algorithm with staff at THETA prior to subject recruitment. Our team of investigators remained blinded to ensure impartiality in decisions about procedures and analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ODYSSEE-vCHAT (Experimental): ODYSSEE-vCHAT consisted of:
  * Automated digital counselling resources (educational pages, videos, tools, and trackers)
  * Chatrooms available 24/7
  * Weekly 30-minute webcasts led by a healthcare professional or patient representative
  Each aspect was informed by a rotating schedule of 7 weekly self-care themes. Webcasts were recorded and streamed to our private YouTube channel, and associated hyperlinks were shared on the program. Subjects had the option of submitting photographs depicting heart-healthy lifestyles and activities (with no identifying, sensitive, or personal information) to the Gallery Wall.
  Subjects were invited by email to access the resources available to them. They logged on to the program using password-protected personal accounts. Each participant's total number of logins and login time (with timestamps) were recorded. Assessments occurred online at baseline, months 4, 8, and 12, and trial completion (median = 8.5 months, range = 2 to 15 months).
  Interventions: Behavioral: ODYSSEE-vCHAT
- eUC (No Intervention): eUC provided educational HF self-care resources that are available to the public on professional heart health websites (e.g., Heart Failure Society of Canada, American Heart Association, European Society of Cardiology, Health Canada). Patients were provided with unlimited access to these resources. Subjects were invited by weekly emails to partake in these resources. Self-reported assessments are administered at baseline, months 4, 8, and 12, and trial completion (median = 8.5 months, range = 2 to 15 months).

INTERVENTIONS:
Behavioral: ODYSSEE-vCHAT — Automated digital counselling program with social network support
  Arms: ODYSSEE-vCHAT

SUMMARY:
INTRODUCTION

Psychological distress and reduced quality of life are prevalent within the heart failure (HF) population. The 1-year rehospitalization (40%) and 5-year mortality (45% for women and 60% for men) rates are high. International task force committees report that medical therapy combined with counselling for HF self-care optimizes clinical outcomes.

HYPOTHESES

At trial completion (median = 8.5 months, range = 2 to 15 months), ODYSSEE-vCHAT versus enhanced usual care (eUC) is predicted to reduce morbidity and mortality rates. Greater engagement with the digital program is also predicted to be linked with improved self-reported mental and physical health at months 4, 8, and 12 and trial completion.

RECRUITMENT

HF patients who are at least 18 years old were recruited from the University Health Network (UHN), Sunnybrook Hospital, Mount Sinai Hospital, and the community. Accrual of the sample (N = 61) occurred over 13 months.

DESIGN

ODYSSEE-vCHAT is a double-arm, parallel-group, randomized, controlled (real-world) pilot trial with assessments at baseline, months 4, 8, and 12, and trial completion (median = 8.5 months, range = 2 to 15 months). It is a single-blind trial, with research personnel blinded (excluding the research coordinator). All patients were provided with free access to their respective digital intervention, ODYSSEE-vCHAT or eUC. Subjects were invited by weekly emails to participate in the resources available to their group. eUC patients were provided with access to educational materials for HF self-care that are available to the public on professional heart health websites. Participation in supplementary programs that provide HF self-care education was not restricted, rather it was monitored by self-report during assessments and will be statistically controlled for during outcome assessments.

ANALYSIS

Separate generalized linear models (GLMs) will evaluate ODYSSEE-vCHAT versus eUC for primary and secondary outcomes. GLMs will be adjusted for baseline assessments and potential covariates. Interactions between treatment arm and gender will be examined for each outcome, using Bonferroni post-hoc comparisons for relevant subgroups. Significance in all tests will be p < 0.05, 2-sided.

DETAILED DESCRIPTION:
BACKGROUND

HF is a progressive clinical syndrome in which the heart is unable to pump oxygenated blood to meet the body's metabolic demands during exercise or at rest. At 55 years, the lifetime risk for HF is 29% for women and 33% for men. HF is a major cause of psychological distress and reduced quality of life. The 1-year rehospitalization rate is 40%. The 5-year mortality rate is 45% and 60% for women and men, respectively.

The incidence of cardiovascular mortality decreases with incremental adherence to self-care. Improvement in HF self-care also predicts greater quality of life at 12 months. However, in the absence of intervention, only 9-36% of HF patients have moderate to high adherence to these behaviours. Barriers to self-care include poor health literacy and social isolation, which are present in 39% and 25% of HF patients, respectively. These barriers are associated with depressed mood and low motivation, both of which increase the risk for poor clinical outcomes.

Home-based telehealth programs such as the present ODYSSEE-vCHAT digital initiative are changing practice standards for outpatient medical care. A telehealth program of social network support that is integrated with automated digital counselling is central to this proposal. This approach has demonstrated potential to improve overall wellbeing and sustain positive behavioural changes through information sharing, structured presentations, and role modelling.

RATIONALE

Task force statements advocate for digital interventions that are patient-centred, scalable, and can improve clinical outcomes while reducing healthcare costs. Furthermore, the development of home-based telehealth programs such as ODYSSEE-vCHAT is consistent with guidelines for COVID-19 prevention. Furthermore, integrating a social network intervention with an automated (scalable), evidence-based digital program for HF self-care is likely to optimize therapeutic benefits. A digital social network initiative is central to this trial because of its potential to (i) sustain patient engagement with HF self-care resources, (ii) promote self-care learning and positive role modelling through information sharing and structured presentations, and (iii) improve quality of life and health literacy while reducing perceived social isolation.

HYPOTHESES

The primary hypothesis is that ODYSSEE-vCHAT versus eUC will reduce the risk for a composite index of incident all-cause mortality, all-cause emergency department (ED) visits, and HF-related hospitalization (based on linkage to health administrative a data base) at trial completion (median = 8.5 months, range = 2 to 15 months).

The secondary hypothesis is that engagement with HF self-care resources [defined by (i) sum logon minutes, (ii) sum logons, and (iii) number of logon days prior to a logon lapse ≥ 2 months] at months 4, 8, and 12 and trial completion (range = 2 to 15 months) will be independently associated with the following outcomes:

* Health-related quality of life
* Adherence to HF self-care
* Engagement in activities for living well
* Overall mental health
* Health literacy
* Active involvement in medical care
* Perceived social support
* Depression
* Anxiety
* Loneliness
* Use of alcohol, cigarettes, and cannabis

POTENTIAL RISKS

Participants may have experienced discomfort with the following:

* Responding to items in the assessments that are considered personal
* Using ODYSSEE-vCHAT because they are not familiar with the software
* Verbally contributing to the discussion segments of the webcasts as their voice would be recorded
* Submitting an audio or video response to the webcasts because they would no longer be an anonymous participant (audio or video comments may also be used for research and educational purposes in the public domain)

SAFETY PARAMETERS

Refusals to respond to any item(s) posed in the questionnaire packages were accommodated.

Video tutorials on how to use ODYSSEE-vCHAT were provided. Assistance over the telephone was offered when required.

During webcasts, visual input from patients remained disabled to protect their identification. If participants preferred to contribute to the discussion without speaking, they were encouraged to use the chat feature on Zoom instead. Comments written in the chat were not included in the recording of the session.

Participants' audio or video comments were censored for inappropriate comments pertaining to violence, sexual content, coarse language, etc. In regards to videos that were selected for presentation to other participants in the trial, or to the public, patients were notified so that they have an opportunity to grant or withhold their permission for this use of their video.

Social network chatrooms are HIPPA compliant and moderated by three levels of content filtering to ensure that posts meet conventional standards of ethical conduct. Level 1 was a search algorithm that is automatically updated with banned word lists. Level 2 was carried by patient volunteers through self-report. Level 3 is performed by research assistants.

Finally, subjects in the intervention arm were offered an opportunity to send the unblinded research coordinator photographs via email which depict heart-healthy lifestyles. Patients were asked not to include any identifying, sensitive, or personal information (e.g., faces, family members, personal health information, etc.) in the photographs, which would be shared with other participants to encourage social interaction. Participants were informed that they could contact the research team at any time to have their photo submissions withdrawn.

STATISTICAL PLAN

Primary outcome:

At trial completion (median = 8.5 months, range = 2 to 15 months), a time-to-event analysis will be conducted using a multivariable Cox Proportional Hazards model to evaluate if ODYSSEE-vCHAT versus eUC reduced the composite endpoint. Potential confounders will be selected using forward (p < 0.05) and backward (p < 0.10) stepwise selection.

Secondary outcomes:

GLMs will evaluate if ODYSSEE-vCHAT versus eUC evokes greater program adherence at months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months), adjusting for potential baseline confounders. The GLM will be repeated using sum logons as the dependent variable. A multivariable Poisson model will evaluate whether ODYSSEE-vCHAT versus eUC is associated with greater duration of engagement, adjusting for potential confounding variables. Separate GLMs will evaluate if ODYSSEE-vCHAT versus eUC improves self-reported outcomes at months 4, 8, and 12 and trial completion, adjusting for endpoints at baseline and potential baseline covariates. Clinical interpretation for health-related quality of life will be based on a group difference of greater than or equal to 5 points. Bonferroni post-hoc tests will be used to assess interactions for relevant groups. Significance in all tests will be p < 0.05, 2-sided.

Exploratory outcomes:

Separate analyses will be conducted for gender. The Cox Proportional Hazards Model or competing risk models will be used for HF-specific endpoints of mortality, hospitalization, and ED visits, separately and collectively.

DEVIATIONS FROM STATISTICAL PLAN

A need to deviate from the statistical plan was not expected as it involves exploratory analyses. Nevertheless, the Statistical Analysis and Methodology Committee was consulted regularly throughout the trial. Any unplanned analyses will be adjusted using the Bonferroni procedure.

SAMPLE SIZE

Researchers recently reported a reduction over 12 months in a composite index score of all-cause mortality and hospitalization for telehealth support (50.6%) versus usual care (59.3%), p = 0.01. This yielded a sample estimate of 142. Using a 14.7% adjustment rate (142 × 1.147) for withdrawal or attrition based on values obtained from CHF-CePPORT (6.5% of patients withdrew and 8.2% were lost to follow-up), the final sample size estimate was 162, with a type 1 error of 5% and a power of 80%. However, the accrued sample size was N = 61.

COMPLIANCE

Attendance for assessments was facilitated by telephone and email reminders if a participant fails to complete an assessment within 5 to 7 days of receiving the initial invitation.

WITHDRAWAL

Adverse events such as an unforeseen mental health crisis may have affected a patient's ability to participate in this trial. In cases of patient withdrawal, all data up to this point pertaining to the patient will be used for outcome analyses. The Steering Committee were responsible for reviewing how and whether the subject should be replaced in the trial. The referring cardiologist would have been alerted about the withdrawal.

CRITERIA FOR TRIAL TERMINATION

The ODYSSEE-vCHAT trial would have been terminated prematurely in the event of a recurrent adverse event that was related to our trial procedures or content.

QUALITY CONTROL AND ASSURANCE

The Data Review or Monitoring Committee ensured that the trial met an appropriate standard for data quality control. The Steering Committee adjudicated primary and secondary outcomes, as well as reviewed and advised the team about the trial's progress, protocol compliance, and any adverse incidents.

CONSENT

Cardiologists and their nursing staff in participating outpatient clinics identified patients who met trial criteria and obtained verbal consent to be approached by the research team. Research personnel either approached the potential participant in the clinic or entered electronic patient records to obtain their contact information. Informed consent was obtained in person or virtually.

This trial was advertised to HF patients on patient education websites, on posters in participating outpatient clinics, and through mass emails. Patients who contacted the research team through advertising were sent our Referral Form via email to be completed and returned via email by their physician. The Referral Form screened potential participants based on the inclusion and exclusion criteria. Potential participants who qualified for the trial were then directed through the consenting process virtually.

DATA STORAGE

All data is stored on secure servers within the UHN digital environment and will remain there for at least 10 years after trial completion.

Data will be available from the corresponding author pending approval of research ethics boards of participating institutions and on reasonable request received from qualified researchers trained in human subject confidentiality protocols.

PRIVACY AND CONFIDENTIALITY

Subjects are issued a tracking number when data involving identifying information is transmitted for analysis. Subject anonymity and confidentiality has been preserved. Only aggregate data will be published.

All research personnel have signed an employee confidentiality agreement ensuring that confidential information is not disclosed to any other person or entity. All source documents containing personal identifiers are stored in filing cabinets under lock and key. The database is stored electronically on the firewall-protected server, making it inaccessible externally. Access to the room containing the research file server is restricted to designated persons who are employed by the Behavioural Cardiology Research Unit at the UHN.

Discussion of the trial with persons outside the research team will never reveal personal identifiers of participants. All access to data is denied to persons outside the research team. Data transmission occurs via encrypted storage material over the Internet.

ELIGIBILITY:
Inclusion criteria:

* Biological males and females who are at least 18 years old and diagnosed with HF with reduced, mid-range, or preserved ejection fraction corresponding to the New York Heart Association Classes 2 to 4 (NYHA II-IV) for 3 or more months prior to enrollment
* Reduced (less than or equal to 40%), mid-range (41 to 49%), or preserved (equal to or greater than 50%) left ventricular ejection fraction, with documentation by ventriculography or quantitative echocardiography (these data are readily available as per the standard of care)
* No worsening of HF for 1 month prior to recruitment, as determined by a referring physician
* Receiving medical treatment in compliance with the Canadian Cardiovascular Society's guideline-directed therapy for at least 1 month prior to enrollment
* Oral and written comprehension of English
* Personal access to an email address, a computer, and the Internet
* Informed written consent

Exclusion criteria:

* Scheduled for advanced surgical therapy (e.g., heart transplantation or implantation of a left ventricular assistive device) within 3 months of enrollment
* Record of significant comorbidities at enrollment that is expected to prohibit full participation (e.g., dementia, psychosis, or severe depression)
* HF secondary to uncorrected valvular cardiomyopathy, predominant right-sided HF, or a non-cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Composite index of incident all-cause mortality, all-cause ED visits, and HF-related hospitalization | Trial completion (median = 8.5 months, range = 2 to 15 months)
  The primary goal of the trial is to evaluate whether use of ODYSSEE-vCHAT versus eUC reduces the risk for a composite index of incident all-cause mortality, all-cause ED visits, and HF-related hospitalization. This data will be collected using the Ontario population-based databases at the Institute for the Clinical Evaluative Sciences (ICES). Data for patients will be linked to ICES databases via Ontario Health Insurance Plan (OHIP) number, first and last name, and date of birth using deterministic/probabilistic linkage (patient unique IKN number).

SECONDARY OUTCOMES:
Incidence of all-cause mortality | Trial completion (median = 8.5 months, range = 2 to 15 months)
  This data will be collected using ICES. Data for patients will be linked to ICES databases via OHIP number, first and last name, and date of birth using deterministic/probabilistic linkage (patient unique IKN number).
Incidence of all-cause ED visits | Trial completion (median = 8.5 months, range = 2 to 15 months)
  This data will be collected using ICES. Data for patients will be linked to ICES databases via OHIP number, first and last name, and date of birth using deterministic/probabilistic linkage (patient unique IKN number).
Incidence of HF-related hospitalization | Trial completion (median = 8.5 months, range = 2 to 15 months)
  This data will be collected using ICES. Data for patients will be linked to ICES databases via OHIP number, first and last name, and date of birth using deterministic/probabilistic linkage (patient unique IKN number).
Engagement with HF self-care resources | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Total number of logon minutes, total number of logons, and number of logon days prior to a logon lapse greater than or equal to 2 months
Self-reported health-related quality of life | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  12-Item Kansas City Cardiomyopathy Questionnaire (KCCQ-12), with clinical interpretation based on a group difference of greater than or equal to 5 points
Adherence to heart failure self-care behaviours | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  9-Item European Heart Failure Self-care Behaviour scale (EHFScB-9)
Self-reported engagement in activities for living well | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Evaluation of Goal-Directed Behaviours to Promote Well-Being and Health (EUROIA), developed by the principal investigator
Self-reported overall mental health | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Mental Component Summary (MCS) of the 36-Item Short-Form survey (SF-36)
Self-reported depression | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  9-Item Patient Health Questionnaire (PHQ-9)
Self-reported anxiety | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  7-Item Generalized Anxiety Disorder instrument (GAD-7)
Self-reported loneliness | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  6-Item Revised UCLA Loneliness Scale (RULS-6)
Self-reported psychological wellbeing | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Flourishing Scale (FS)
Self-reported involvement in medical care | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  6-Item Self-Efficacy for Managing Chronic Disease instrument (SEMCD-6)
Self-reported health literacy | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Developed by the principal investigator
Self-reported physical wellbeing | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ)
Self-reported perceived social support | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  ENRICHD Social Support Instrument (ESSI)
Self-reported alcohol, nicotine, and cannabis use | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)

OTHER OUTCOMES:
Gender interactions | Months 4, 8, and 12 and trial completion (median = 8.5 months, range = 2 to 15 months)
  Exploratory analyses will be conducted for gender categories represented by participants (male, female, gender fluid or non-binary, and not specified).

CONTACTS AND LOCATIONS:
Overall Officials: Rob P Nolan, PhD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - University Health Network, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutledge T, Reis VA, Linke SE, Greenberg BH, Mills PJ. Depression in heart failure a meta-analytic review of prevalence, intervention effects, and associations with clinical outcomes. J Am Coll Cardiol. 2006 Oct 17;48(8):1527-37. doi: 10.1016/j.jacc.2006.06.055. Epub 2006 Sep 26. PMID 17045884
- [Background] Dekker RL. Patient perspectives about depressive symptoms in heart failure: a review of the qualitative literature. J Cardiovasc Nurs. 2014 Jan-Feb;29(1):E9-15. doi: 10.1097/JCN.0b013e318273a5d6. PMID 23151836
- [Background] Lee KS, Lennie TA, Wu JR, Biddle MJ, Moser DK. Depressive symptoms, health-related quality of life, and cardiac event-free survival in patients with heart failure: a mediation analysis. Qual Life Res. 2014 Aug;23(6):1869-76. doi: 10.1007/s11136-014-0636-5. Epub 2014 Feb 1. PMID 24488573
- [Background] Lee DS, Johansen H, Gong Y, Hall RE, Tu JV, Cox JL; Canadian Cardiovascular Outcomes Research Team. Regional outcomes of heart failure in Canada. Can J Cardiol. 2004 May 1;20(6):599-607. PMID 15152289
- [Background] Malcom J, Arnold O, Howlett JG, Ducharme A, Ezekowitz JA, Gardner M, Giannetti N, Haddad H, Heckman GA, Isaac D, Jong P, Liu P, Mann E, McKelvie RS, Moe GW, Svendsen AM, Tsuyuki RT, O'Halloran K, Ross HJ, Sequeira EJ, White M; Canadian Cardiovascular Society. Canadian Cardiovascular Society Consensus Conference guidelines on heart failure--2008 update: best practices for the transition of care of heart failure patients, and the recognition, investigation and treatment of cardiomyopathies. Can J Cardiol. 2008 Jan;24(1):21-40. doi: 10.1016/s0828-282x(08)70545-2. PMID 18209766
- [Background] Ezekowitz JA, O'Meara E, McDonald MA, Abrams H, Chan M, Ducharme A, Giannetti N, Grzeslo A, Hamilton PG, Heckman GA, Howlett JG, Koshman SL, Lepage S, McKelvie RS, Moe GW, Rajda M, Swiggum E, Virani SA, Zieroth S, Al-Hesayen A, Cohen-Solal A, D'Astous M, De S, Estrella-Holder E, Fremes S, Green L, Haddad H, Harkness K, Hernandez AF, Kouz S, LeBlanc MH, Masoudi FA, Ross HJ, Roussin A, Sussex B. 2017 Comprehensive Update of the Canadian Cardiovascular Society Guidelines for the Management of Heart Failure. Can J Cardiol. 2017 Nov;33(11):1342-1433. doi: 10.1016/j.cjca.2017.08.022. Epub 2017 Sep 6. PMID 29111106
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Bleumink GS, Knetsch AM, Sturkenboom MC, Straus SM, Hofman A, Deckers JW, Witteman JC, Stricker BH. Quantifying the heart failure epidemic: prevalence, incidence rate, lifetime risk and prognosis of heart failure The Rotterdam Study. Eur Heart J. 2004 Sep;25(18):1614-9. doi: 10.1016/j.ehj.2004.06.038. PMID 15351160
- [Background] Bramley TJ, Gerbino PP, Nightengale BS, Frech-Tamas F. Relationship of blood pressure control to adherence with antihypertensive monotherapy in 13 managed care organizations. J Manag Care Pharm. 2006 Apr;12(3):239-45. doi: 10.18553/jmcp.2006.12.3.239. PMID 16623608
- [Background] Granger BB, Swedberg K, Ekman I, Granger CB, Olofsson B, McMurray JJ, Yusuf S, Michelson EL, Pfeffer MA; CHARM investigators. Adherence to candesartan and placebo and outcomes in chronic heart failure in the CHARM programme: double-blind, randomised, controlled clinical trial. Lancet. 2005 Dec 10;366(9502):2005-11. doi: 10.1016/S0140-6736(05)67760-4. PMID 16338449
- [Background] Khaw KT, Wareham N, Bingham S, Welch A, Luben R, Day N. Combined impact of health behaviours and mortality in men and women: the EPIC-Norfolk prospective population study. PLoS Med. 2008 Jan 8;5(1):e12. doi: 10.1371/journal.pmed.0050012. PMID 18184033
- [Background] Rasmussen JN, Chong A, Alter DA. Relationship between adherence to evidence-based pharmacotherapy and long-term mortality after acute myocardial infarction. JAMA. 2007 Jan 10;297(2):177-86. doi: 10.1001/jama.297.2.177. PMID 17213401
- [Background] Simpson SH, Eurich DT, Majumdar SR, Padwal RS, Tsuyuki RT, Varney J, Johnson JA. A meta-analysis of the association between adherence to drug therapy and mortality. BMJ. 2006 Jul 1;333(7557):15. doi: 10.1136/bmj.38875.675486.55. Epub 2006 Jun 21. PMID 16790458
- [Background] Musekamp G, Schuler M, Seekatz B, Bengel J, Faller H, Meng K. Does improvement in self-management skills predict improvement in quality of life and depressive symptoms? A prospective study in patients with heart failure up to one year after self-management education. BMC Cardiovasc Disord. 2017 Feb 15;17(1):51. doi: 10.1186/s12872-017-0486-5. PMID 28196523
- [Background] Evangelista LS, Shinnick MA. What do we know about adherence and self-care? J Cardiovasc Nurs. 2008 May-Jun;23(3):250-7. doi: 10.1097/01.JCN.0000317428.98844.4d. PMID 18437067
- [Background] Marti CN, Georgiopoulou VV, Giamouzis G, Cole RT, Deka A, Tang WH, Dunbar SB, Smith AL, Kalogeropoulos AP, Butler J. Patient-reported selective adherence to heart failure self-care recommendations: a prospective cohort study: the Atlanta Cardiomyopathy Consortium. Congest Heart Fail. 2013 Jan-Feb;19(1):16-24. doi: 10.1111/j.1751-7133.2012.00308.x. Epub 2012 Sep 9. PMID 22958604
- [Background] Cajita MI, Cajita TR, Han HR. Health Literacy and Heart Failure: A Systematic Review. J Cardiovasc Nurs. 2016 Mar-Apr;31(2):121-30. doi: 10.1097/JCN.0000000000000229. PMID 25569150
- [Background] Manemann SM, Chamberlain AM, Roger VL, Griffin JM, Boyd CM, Cudjoe TKM, Jensen D, Weston SA, Fabbri M, Jiang R, Finney Rutten LJ. Perceived Social Isolation and Outcomes in Patients With Heart Failure. J Am Heart Assoc. 2018 May 23;7(11):e008069. doi: 10.1161/JAHA.117.008069. PMID 29794038
- [Background] Zou H, Chen Y, Fang W, Zhang Y, Fan X. The mediation effect of health literacy between subjective social status and depressive symptoms in patients with heart failure. J Psychosom Res. 2016 Dec;91:33-39. doi: 10.1016/j.jpsychores.2016.10.006. Epub 2016 Oct 19. PMID 27894460
- [Background] Matsuoka S, Kato N, Kayane T, Yamada M, Koizumi M, Ikegame T, Tsuchihashi-Makaya M. Development and Validation of a Heart Failure-Specific Health Literacy Scale. J Cardiovasc Nurs. 2016 Mar-Apr;31(2):131-9. doi: 10.1097/JCN.0000000000000226. PMID 26049813
- [Background] Zou H, Chen Y, Fang W, Zhang Y, Fan X. Identification of factors associated with self-care behaviors using the COM-B model in patients with chronic heart failure. Eur J Cardiovasc Nurs. 2017 Aug;16(6):530-538. doi: 10.1177/1474515117695722. Epub 2017 Feb 1. PMID 28756696
- [Background] Bauer LK, Caro MA, Beach SR, Mastromauro CA, Lenihan E, Januzzi JL, Huffman JC. Effects of depression and anxiety improvement on adherence to medication and health behaviors in recently hospitalized cardiac patients. Am J Cardiol. 2012 May 1;109(9):1266-71. doi: 10.1016/j.amjcard.2011.12.017. Epub 2012 Feb 9. PMID 22325974
- [Background] Tierney S, Mamas M, Woods S, Rutter MK, Gibson M, Neyses L, Deaton C. What strategies are effective for exercise adherence in heart failure? A systematic review of controlled studies. Heart Fail Rev. 2012 Jan;17(1):107-15. doi: 10.1007/s10741-011-9252-4. PMID 21567221
- [Background] Moraska AR, Chamberlain AM, Shah ND, Vickers KS, Rummans TA, Dunlay SM, Spertus JA, Weston SA, McNallan SM, Redfield MM, Roger VL. Depression, healthcare utilization, and death in heart failure: a community study. Circ Heart Fail. 2013 May;6(3):387-94. doi: 10.1161/CIRCHEARTFAILURE.112.000118. Epub 2013 Mar 19. PMID 23512984
- [Background] Daniel H, Sulmasy LS; Health and Public Policy Committee of the American College of Physicians. Policy recommendations to guide the use of telemedicine in primary care settings: an American College of Physicians position paper. Ann Intern Med. 2015 Nov 17;163(10):787-9. doi: 10.7326/M15-0498. Epub 2015 Sep 8. PMID 26344925
- [Background] Cowie MR, Bax J, Bruining N, Cleland JG, Koehler F, Malik M, Pinto F, van der Velde E, Vardas P. e-Health: a position statement of the European Society of Cardiology. Eur Heart J. 2016 Jan 1;37(1):63-6. doi: 10.1093/eurheartj/ehv416. Epub 2015 Aug 24. No abstract available. PMID 26303835
- [Background] Eapen ZJ, Turakhia MP, McConnell MV, Graham G, Dunn P, Tiner C, Rich C, Harrington RA, Peterson ED, Wayte P. Defining a Mobile Health Roadmap for Cardiovascular Health and Disease. J Am Heart Assoc. 2016 Jul 12;5(7):e003119. doi: 10.1161/JAHA.115.003119. No abstract available. PMID 27405809
- [Background] Bhavnani SP, Parakh K, Atreja A, Druz R, Graham GN, Hayek SS, Krumholz HM, Maddox TM, Majmudar MD, Rumsfeld JS, Shah BR. 2017 Roadmap for Innovation-ACC Health Policy Statement on Healthcare Transformation in the Era of Digital Health, Big Data, and Precision Health: A Report of the American College of Cardiology Task Force on Health Policy Statements and Systems of Care. J Am Coll Cardiol. 2017 Nov 28;70(21):2696-2718. doi: 10.1016/j.jacc.2017.10.018. No abstract available. PMID 29169478
- [Background] Stogios N, Kaur B, Huszti E, Vasanthan J, Nolan RP. Advancing Digital Health Interventions as a Clinically Applied Science for Blood Pressure Reduction: A Systematic Review and Meta-analysis. Can J Cardiol. 2020 May;36(5):764-774. doi: 10.1016/j.cjca.2019.11.010. Epub 2019 Nov 15. PMID 32249065
- [Background] Wu RC, Delgado D, Costigan J, Ross H, MacIver J. Pilot study of an Internet patient-physician communication tool for heart failure disease management. World Hosp Health Serv. 2006;42(3):32-8. PMID 17249472
- [Background] Sakakibara BM, Ross E, Arthur G, Brown-Ganzert L, Petrin S, Sedlak T, Lear SA. Using Mobile-Health to Connect Women with Cardiovascular Disease and Improve Self-Management. Telemed J E Health. 2017 Mar;23(3):233-239. doi: 10.1089/tmj.2016.0133. Epub 2016 Sep 13. PMID 27623231
- [Background] van Woudenberg TJ, Simoski B, Fernandes de Mello Araujo E, Bevelander KE, Burk WJ, Smit CR, Buijs L, Klein M, Buijzen M. Identifying Influence Agents That Promote Physical Activity Through the Simulation of Social Network Interventions: Agent-Based Modeling Study. J Med Internet Res. 2019 Aug 5;21(8):e12914. doi: 10.2196/12914. PMID 31381504
- [Background] Chung ML, Moser DK, Lennie TA, Frazier SK. Perceived social support predicted quality of life in patients with heart failure, but the effect is mediated by depressive symptoms. Qual Life Res. 2013 Sep;22(7):1555-63. doi: 10.1007/s11136-012-0294-4. Epub 2012 Oct 18. PMID 23076798
- [Background] Trinacty M, Farrell B, Schindel TJ, Sunstrum L, Dolovich L, Kennie N, Russell G, Waite N. Learning and networking: utilization of a primary care listserv by pharmacists. Can J Hosp Pharm. 2014 Sep;67(5):343-52. doi: 10.4212/cjhp.v67i5.1388. PMID 25364016
- [Background] Seidel RL, Jalilvand A, Kunjummen J, Gilliland L, Duszak R Jr. Radiologists and Social Media: Do Not Forget About Facebook. J Am Coll Radiol. 2018 Jan;15(1 Pt B):224-228. doi: 10.1016/j.jacr.2017.09.013. Epub 2017 Nov 11. PMID 29132999
- [Background] Gomez-Pardo E, Fernandez-Alvira JM, Vilanova M, Haro D, Martinez R, Carvajal I, Carral V, Rodriguez C, de Miguel M, Bodega P, Santos-Beneit G, Penalvo JL, Marina I, Perez-Farinos N, Dal Re M, Villar C, Robledo T, Vedanthan R, Bansilal S, Fuster V. A Comprehensive Lifestyle Peer Group-Based Intervention on Cardiovascular Risk Factors: The Randomized Controlled Fifty-Fifty Program. J Am Coll Cardiol. 2016 Feb 9;67(5):476-85. doi: 10.1016/j.jacc.2015.10.033. Epub 2015 Nov 9. PMID 26562047
- [Background] Wu JR, Frazier SK, Rayens MK, Lennie TA, Chung ML, Moser DK. Medication adherence, social support, and event-free survival in patients with heart failure. Health Psychol. 2013 Jun;32(6):637-46. doi: 10.1037/a0028527. Epub 2012 Jul 2. PMID 22746258
- [Background] Rodriguez-Artalejo F, Guallar-Castillon P, Herrera MC, Otero CM, Chiva MO, Ochoa CC, Banegas JR, Pascual CR. Social network as a predictor of hospital readmission and mortality among older patients with heart failure. J Card Fail. 2006 Oct;12(8):621-7. doi: 10.1016/j.cardfail.2006.06.471. PMID 17045181
- [Background] Bonniface L, Green L. Finding a new kind of knowledge on the HeartNET website. Health Info Libr J. 2007 Dec;24 Suppl 1:67-76. doi: 10.1111/j.1471-1842.2007.00742.x. PMID 18005296
- [Background] Lau AY, Dunn A, Mortimer N, Proudfoot J, Andrews A, Liaw ST, Crimmins J, Arguel A, Coiera E. Consumers' online social network topologies and health behaviours. Stud Health Technol Inform. 2013;192:77-81. PMID 23920519
- [Background] Gammon D, Strand M, Eng LS, Borosund E, Varsi C, Ruland C. Shifting Practices Toward Recovery-Oriented Care Through an E-Recovery Portal in Community Mental Health Care: A Mixed-Methods Exploratory Study. J Med Internet Res. 2017 May 2;19(5):e145. doi: 10.2196/jmir.7524. PMID 28465277
- [Background] Toukhsati SR, Driscoll A, Hare DL. Patient Self-management in Chronic Heart Failure - Establishing Concordance Between Guidelines and Practice. Card Fail Rev. 2015 Oct;1(2):128-131. doi: 10.15420/cfr.2015.1.2.128. PMID 28785446
- [Background] Nolan RP, Payne AY, Ross H, White M, D'Antono B, Chan S, Barr SI, Gwadry-Sridhar F, Nigam A, Perreault S, Farkouh M, McDonald M, Goodman J, Thomas S, Zieroth S, Isaac D, Oh P, Rajda M, Chen M, Eysenbach G, Liu S, Zbib A. An Internet-Based Counseling Intervention With Email Reminders that Promotes Self-Care in Adults With Chronic Heart Failure: Randomized Controlled Trial Protocol. JMIR Res Protoc. 2014 Jan 30;3(1):e5. doi: 10.2196/resprot.2957. PMID 24480783
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Vaglio J Jr, Conard M, Poston WS, O'Keefe J, Haddock CK, House J, Spertus JA. Testing the performance of the ENRICHD Social Support Instrument in cardiac patients. Health Qual Life Outcomes. 2004 May 13;2:24. doi: 10.1186/1477-7525-2-24. PMID 15142277
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Wongpakaran N, Wongpakaran T, Pinyopornpanish M, Simcharoen S, Suradom C, Varnado P, Kuntawong P. Development and validation of a 6-item Revised UCLA Loneliness Scale (RULS-6) using Rasch analysis. Br J Health Psychol. 2020 May;25(2):233-256. doi: 10.1111/bjhp.12404. Epub 2020 Jan 30. PMID 31999891
- [Background] Humeniuk R, Ali R, Babor T, Souza-Formigoni ML, de Lacerda RB, Ling W, McRee B, Newcombe D, Pal H, Poznyak V, Simon S, Vendetti J. A randomized controlled trial of a brief intervention for illicit drugs linked to the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) in clients recruited from primary health-care settings in four countries. Addiction. 2012 May;107(5):957-66. doi: 10.1111/j.1360-0443.2011.03740.x. Epub 2012 Feb 28. PMID 22126102
- [Background] Krum H, Forbes A, Yallop J, Driscoll A, Croucher J, Chan B, Clark R, Davidson P, Huynh L, Kasper EK, Hunt D, Egan H, Stewart S, Piterman L, Tonkin A. Telephone support to rural and remote patients with heart failure: the Chronic Heart Failure Assessment by Telephone (CHAT) study. Cardiovasc Ther. 2013 Aug;31(4):230-7. doi: 10.1111/1755-5922.12009. PMID 23061492
- [Background] Nolan RP, Ross HJ, Farkouh ME, Huszti E, Chan S, Toma M, D'Antono B, White M, Thomas S, Barr SI, Perreault S, McDonald M, Zieroth S, Isaac D, Wielgosz A, Mielniczuk LM. Automated E-Counseling for Chronic Heart Failure: CHF-CePPORT Trial. Circ Heart Fail. 2021 Jan;14(1):e007073. doi: 10.1161/CIRCHEARTFAILURE.120.007073. Epub 2021 Jan 19. PMID 33464959
- [Background] Fezza G, Sansone S, Surikova J, Hustzi E, Ross H and Nolan RP. Patient engagement with an e-Counselling platform is enhanced over 12 months in the CHF-CePPORT trial. Can J Cardiol. 2018;10:148-9.
- [Background] Payne AY, Surikova J, Liu S, Ross H, Mechetiuc T, Nolan RP. Usability Testing of an Internet-Based e-Counseling Platform for Adults With Chronic Heart Failure. JMIR Hum Factors. 2015 May 8;2(1):e7. doi: 10.2196/humanfactors.4125. PMID 27026267
- [Background] Spertus J, Peterson E, Conard MW, Heidenreich PA, Krumholz HM, Jones P, McCullough PA, Pina I, Tooley J, Weintraub WS, Rumsfeld JS; Cardiovascular Outcomes Research Consortium. Monitoring clinical changes in patients with heart failure: a comparison of methods. Am Heart J. 2005 Oct;150(4):707-15. doi: 10.1016/j.ahj.2004.12.010. PMID 16209970
- [Background] Jaarsma T, Arestedt KF, Martensson J, Dracup K, Stromberg A. The European Heart Failure Self-care Behaviour scale revised into a nine-item scale (EHFScB-9): a reliable and valid international instrument. Eur J Heart Fail. 2009 Jan;11(1):99-105. doi: 10.1093/eurjhf/hfn007. PMID 19147463
- [Derived] Peiris RG, Ross H, Chan CT, Poon S, Auguste BL, Rac VE, Farkouh M, McDonald M, Kaczorowski J, Code J, Duero Posada J, Ong S, Kobulnik J, Tomlinson G, Huszti E, Arcand J, Thomas SG, Akbari A, Maunder R, Grover S, Seto E, Simard A, Pope B, Bains M, McIntyre C, Torbay C, Syed F, Nolan RP. Automated digital counselling with social network support as a novel intervention for patients with heart failure: protocol for randomised controlled trial. BMJ Open. 2022 Sep 5;12(9):e059635. doi: 10.1136/bmjopen-2021-059635. PMID 36691152